CLINICAL TRIAL: NCT06660693
Title: Comparison of Medical RESCUE Strategies for Patients With Steroid-refractory Acute Severe Ulcerative Colitis: an Open-label Randomized Controlled Trial (RESCUE-UC).
Brief Title: Comparison of Medical RESCUE Strategies for Patients With Steroid-refractory Acute Severe Ulcerative Colitis
Acronym: RESCUE UC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Neeraj Narula, Principal Investigator, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESCUE-UC
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: Open-label, pragmatic, multi-centre, randomized control trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upadacitinib (treatment arm) (Active Comparator): Participants will receive Upadacitinib 45mg daily, once a day, for at least five days.
  Interventions: Drug: Upadacitinib Oral Product
- Infliximab (standard care) (No Intervention): Participants will receive standard care, which is Infliximab.

INTERVENTIONS:
Drug: Upadacitinib Oral Product — Upadacitinib oral 45mg once daily.
  Arms: Upadacitinib (treatment arm)

SUMMARY:
This study aims to examine patients with acute severe UC who are refractory to intravenous corticosteroids and determine whether a strategy of using upadacitinib first followed by infliximab in upadacitinib non-responders is non-inferior to conventional management with infliximab only.

DETAILED DESCRIPTION:
In acute hospitalized severe, steroid refractory UC, only two medical rescue therapies have been found efficacious in controlled trials and recommended in management, infliximab and cyclosporine. Due to toxicity and nuance in using cyclosporine, infliximab is by far the most commonly used medical rescue therapy in this setting. There is emerging retrospective and prospective case series data suggesting JAK inhibitors, such as tofacitinib or upadacitinib, could also be used for this patient population. JAK inhibitors offer potential advantages including convenience of oral therapy, efficacy independent of serum albumin levels, and no concern for immunogenicity as is seen with anti-TNFs. They also offer a short half-life and are eliminated by humans within 48 hours of the last dose administered. This could be beneficial, as it may offer a chance to use a JAK inhibitor first and switch to infliximab in patients who do not respond to a JAK inhibitor, as theoretically cumulative immunosuppression should not be as high transitioning from a JAK inhibitor to infliximab, as compared to using JAK inhibitor after infliximab failure since there will still be lots of infliximab present owing to its long half-life. It is unclear how JAK inhibitors compare to our standard of care and where they should be positioned in acute severe UC. This study aims to examine patients with acute severe UC who are refractory to intravenous corticosteroids and determine whether a strategy of using upadacitinib first followed by infliximab in upadacitinib non-responders is non-inferior to conventional management with infliximab only.

ELIGIBILITY:
Inclusion Criteria: Adult (≥ 18 - 64 years) male or non-pregnant, non-lactating female patients with:

* Confirmed diagnosis of UC, based on conventional clinical, endoscopic, and/or histologic criteria
* Admitted to hospital with acute severe flare and refractory to three days of intravenous steroids (at minimum of 40mg methylprednisolone, or equivalent, daily). Refractory is defined using the Oxford criteria at day 3 of steroid therapy: presence of > 8 stools/day or CRP > 45 mg/L
* Will undergo or has already undergone a baseline colonoscopy or flexible sigmoidoscopy while in hospital or in the 4 weeks preceding trial entry, with a baseline MES ≥2 based on locally evaluated endoscopy
* Provided written informed consent
* Subject is willing and able to adhere to study procedures, and describe in the procedures that screening and safety monitoring procedures will be applied as per upadacitinib and infliximab Canadian product monographs

Exclusion Criteria:

* Contraindications to receiving either infliximab or upadacitinib (as per current Canadian product monograph)
* Previously used infliximab or a JAK inhibitor for UC
* Patients > 65 years of age
* Pregnant or breastfeeding
* Women of reproductive potential who are unwilling to agree to using effective contraception during treatment and 4 weeks following the final dose of upadacitinib
* Concurrent Clostridium difficile, other gastrointestinal infection, or other active systemic or localized infection which would preclude treatment with systemically acting biologic or small molecule therapy
* Patients with symptoms of thrombosis, or confirmed venous or arterial thromboembolism
* Active TB (patients should be tested for TB prior to upadacitinib or infliximab treatment)
* HBV/HCV positive
* Untreated malignancy or ongoing treatment for malignancy
* Concomitant treatment with strong CYP3A4 inhibitors or inducers
* Severe hepatic impairment
* Severe renal impairment (CrCl < 30 ml/min)
* Patients who have received live vaccines in the 28 days prior to study entry.
* Patients with moderate or severe (NYHA Class III/IV) congestive heart failure.
* Patients with a history of hypersensitivity to infliximab, to other murine proteins, or to any of the excipients.
* Patients who are hypersensitive to upadacitinib or to any ingredient in the formulation, including any non-medicinal ingredient, or component of the container.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Measure treatment success of upadacitinib vs standard care. | 16 weeks
  The primary objective of this study is to evaluate whether treatment success in ASUC patients in patients treated with strategy U is non-inferior to strategy C after 16 weeks of initiating therapeutic management.

CONTACTS AND LOCATIONS:
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada